CLINICAL TRIAL: NCT05502458
Title: Effect of Propofol and Desflurane on Nucleic Acid of Liver Circulating Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fang Jun, clinical professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-09-01
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma; Desflurane Adverse Reaction; Propofol Adverse Reaction; Circulating Tumor Cells
Keywords: Desflurane; HCC; propofol; CTC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating | interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Propofol general anesthesia group (P group) : intravenous propofol infusion was slowly pushed until consciousness disappeared, and then anesthesia was maintained at 4-8 mg/kg/h.
  In the general anesthesia group with desflurane (group D), intravenous propofol infusion was slowly pushed until consciousness disappeared, and then anesthesia was maintained with 4-6% desflurane
Who Masked: Participant, Care Provider
Masking Description: By statistical professionals using SAS software on the computer, according to the propofol group and halothane group the proportion of 1:1, to patients by ASA classification, disease category, coexist, the condition of the body after stratified according to stratified random methods such as random coding, in this study, each participant will be according to the center of the random number sequence into the propofol group and halothane group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propofol (Active Comparator): propofol（50ml,1g）,Intravenous propofol infusion was slowly pushed until loss of consciousness, and anesthesia was maintained at 4-8 mg/kg/h
  Interventions: Drug: Propofol
- desflurane (Active Comparator): In the general anesthesia group with desflurane( 240ml), intravenous propofol infusion was slowly pushed until consciousness disappeared, and then anesthesia was maintained with 4-6% desflurane
  Interventions: Drug: Desﬂurane

INTERVENTIONS:
Drug: Desﬂurane — Propofol general anesthesia group (P group) : intravenous propofol infusion was slowly pushed until consciousness disappeared, and then anesthesia was maintained at 4-8 mg/kg/h. In the general anesthesia group with desflurane (group D), intravenous propofol infusion was slowly pushed until consciousness disappeared, and then anesthesia was maintained with 4-6% desflurane. The analgesic and muscle relaxant regimens were the same in both groups except for sedative drugs. All patients were treated with no medication before operation, and the operation was completed under endotracheal intubation and general anesthesia. The amount of propofol or desflurane was adjusted according to BIS or MAC values and hemodynamic changes during operation. Add 10mg of rocuronium every half hour. Vasoactive drugs can be used to maintain hemodynamic stability during the operation, and corresponding records should be made
  Other Names: group D
  Arms: desflurane
Drug: Propofol — Propofol general anesthesia group (P group) : intravenous propofol infusion was slowly pushed until consciousness disappeared, and then anesthesia was maintained at 4-8 mg/kg/h.
  Other Names: group P
  Arms: propofol

SUMMARY:
To investigate the effects of perioperative anesthetic drugs propofol and desflurane on circulating tumor nucleic acids (CK7, ELF3, EGFR and EphB4 mRNA) in the blood of patients with liver cancer, so as to provide scientific reference for clinical anesthesia in the perioperative treatment of tumor

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most malignant tumors in oncology. Its incidence is increasing, and there is a lack of reliable biomarkers for early diagnosis, prognosis evaluation and efficacy evaluation. There is a pool of tumor molecules derived from primary tumors in the blood circulation, including Circulating tumor proteins, Circulating tumor cells (CTCs), Extracellular vesicles, Evs, Tumor "educated" platelets (TEPs), and Circulating Tumor nucleic acids, known as Circulating Tumor DNA, CtDNA is a Circulating cell-free DNA (ccfDNA). Liquid biopsy is performed to detect tumor molecules from blood circulation. Small RNA (miRNA) and long noncoding RNA (miRNA) in liquid biopsy are detected. Circulating tumor RNA (ctRNA), such as lncRNA, can be used as epigenetic biomarkers to improve the early diagnosis of HCC and to treat patients with early and advanced HCC. Propofol and desflurane, as important anesthesia drugs in perioperative period, have been shown to affect the concentration of circulating nucleic acid in patients. Furong Song found that propofol could inhibit the overexpression of HOXA11-AS, which reversed the inhibitory effect of propofol treatment on HCC cell progression, by promoting the expression of Mir-4458, and had an impact on HCC cell progression . However, Dongmei Wang and their colleagues found that circulating H19 inhibited the effect of propofol in promoting HCC cell apoptosis by upregulating LIMK1 (LIM domain kinase 1) through spongy Mir-520a-3p . Meanwhile, Buschmann and his team found that propofol and desflurane inhibited key cancer-related pathways such as proliferation and migration in colorectal cancer, and found that propofol did not affect the size distribution and protein labeling of circulating vesicles, but could reduce their concentration . Compared with inhaled anesthetics, Bon-Wook Koo found that HCC patients treated with propofol had a lower recurrence rate and a longer average recurrence time than those treated with inhaled anesthetics . Hou-chuan Lai found that compared with desflurane anesthesia regimen, propofol anesthesia regimen significantly improved the survival rate of patients with liver cancer without distant metastasis or local recurrence . Meanwhile, Frederique Hovaguimian found that in nonmetastatic and metastatic breast cancer, the maximum number of circulating tumor cells increased by 36% after sevoflurane inhalation anesthesia and was independently associated with a higher risk of disease recurrence and reduced survival . At this time, the monitoring of circulating tumor cells can represent promising methods, such as the detection of suitable markers of circulating tumor cells, such as Cytokeratin 7 (CK7), E74-like factor 3 (ELF3), Epidermal growth factor receptor (EGFR) and Peripheral blood mononuclear cells, The expression of erythropoietin-producing hepatocellular carcinoma receptor B4 (EphB4) mRNA in PMBCs, In order to better understand the effect of anesthesia on perioperative tumor treatment, this evidence has been supported by domestic and foreign studies . Soo-ho Lee and his colleagues found that CK7-negative liver cancer patients had a higher survival rate than all positive patients [9], which was supported by Xialing Huang and his team . Longbo Zheng found that ELF3 inhibits ZE1 by inhibiting Mir-141-3p, thereby inhibiting E-cadherin in HCC cells and promoting EMT, which is a potential prognostic biomarker and/or therapeutic target for HCC . Zhe Wu found that lncrNA-UBE2R2-AS1 in HCC shows carcinogenic effect through the up-regulation of EGFR by Mir-302b, and can be used as a potential therapeutic target and prognostic biomarker for HCC patients , and this mechanism of action was confirmed by Zhen-Jiang Ma and his research . At the same time, it was found that the expression level of EphB4 was increased in HCC tumor tissues, and the levels of EphB4 and P-JAK2 were positively correlated in samples of HCC patients , while the expression of CIRC-EPHB4 was down-regulated. Circ-ephb4 overexpression inhibited the viability of HCC cells, induced apoptosis, and inhibited cell migration and invasion by inhibiting the expression of hypoxia-inducible factor-1α (HIF-1α) . However, the perioperative effects and molecular mechanisms of propofol and desflurane on circulating tumor nucleic acids in liver cancer are not very clear at present, and further relevant studies are needed to clarify, so as to provide support and guidance for the development of perioperative anesthesia plan and clinical diagnosis of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 to 75
* ASA: I-III
* primary liver cancer (CNLC: Stage I-IIIA)
* undergoing elective hepatectomy

Exclusion Criteria:

* Patients with severe bradycardia (HR < 55bpm)
* patients with severe arrhythmias or cardiac dysfunction (EF < 35%)
* patients with severe respiratory lung disease
* patients with severe liver and kidney insufficiency epilepsy
* patients with severe hyperlipidemia
* patients with a history of malignant hyperthermia
* patients with propofol or desflurane allergy
* patients with history of preoperative chemoradiotherapy
* patients who were on immunosuppressive treatment
* patients with chronic opioid therapy declined to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
The changes of circulating tumor nucleic acids (CK7, ELF3, EGFR and EphB4 mRNA) in peripheral blood of patients with hepatocellular carcinoma after perioperative treatment with propofol and desflurane | Immediately Before induction of anesthesia, Immediately before skinning after induction of anesthesia, during operation, PACU at the end of operation, and on the 7th day after operation
  Circulating tumor nucleic acid (CK7, ELF3, EGFR, and EphB4 mRNA) concentrations were determined by real-time RT-PCR in Applied Biosystems 7500 (Foster City, CA, USA) using SYBR® Premix Ex TaqTM II (Po, Otsu, Japan). Sequence of primers designed as previously described. Total mRNA was normalized to GAPDH and relative mRNA expression of the sample by calculating 2- δδCT, and differential expression of the sample was defined as upregulation when the cutoff value was set to 2x

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer hospital, Hangzhou, Zhejiang, China